CLINICAL TRIAL: NCT01927367
Title: Integrated Management Program Advancing Community Treatment of Atrial Fibrillation (IMPACT-AF)
Brief Title: Integrated Management Program Advancing Community Treatment of Atrial Fibrillation
Acronym: IMPACT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jafna L Cox (Other)
Collaborators: McMaster University (Other); Population Health Research Institute (Other); St. Joseph's Healthcare Hamilton (Other); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Jafna L Cox, Staff Cardiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMPACT-AF-2013
Record Dates: First submitted 2013-08-20; First posted 2013-08-22 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
Keywords: Clinical Decision Support System; Primary Health Care; Clinical Practice Guidelines
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical Decision Support System for AF (Other): Providers randomized to use the Clinical Decision Support System (CDSS, a web-based tool).
  Interventions: Other: Clinical Decision Support System for AF
- Usual Care (No Intervention): Usual Care - providers are not eligible to access / use the CDSS.

INTERVENTIONS:
Other: Clinical Decision Support System for AF — A web-based clinical decision support system, computerizing the Canadian AF clinical guidelines and best-practice approaches, to support primary care providers and patients in optimizing and standardizing AF care.
  Other Names: CDSS
  Arms: Clinical Decision Support System for AF

SUMMARY:
Research Question: Among community-based patients with AF, does providing an integrated Clinical Decision Support System (CDSS) to providers and patients improve process of care and clinical outcomes, and decrease the healthcare costs and resource utilization over 12 months, as compared to usual care?

Intervention: A web-based clinical decision support system, computerizing the Canadian AF clinical guidelines, to support primary care providers and patients in optimizing and standardizing AF care.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common abnormality of cardiac rhythm. It is also a disease of aging, affecting 3% of adults aged > 45 years and 12% of those aged > 75. Individually, AF's rapid and irregular heart beat is most frequently perceived as undesirable palpitations, but more threatening impacts are heart failure, catastrophic stroke and premature death. AF also markedly impairs quality of life.

Although patients with AF are at increased risk of stroke, death and hospitalization, many patients are not benefiting from evidence-informed, best-care strategies. Gaps have been documented in the knowledge, skills and competencies of primary care clinicians concerning the management of AF in Canada. For example, a large proportion of AF patients at moderate to high risk for stroke do not receive guideline recommended thromboprophylaxis; and of those that do, many are not optimally controlled. One Canadian study also found that in patient with known AF and a prior stroke, who were then admitted with a second stroke, 15% were not on any anticoagulation and only 18% were on warfarin and within the therapeutic range. Opportunities certainly exist to enhance the uptake of the Canadian AF Clinical Practice Guideline recommendations and best-care approaches in the primary care setting.

Patients need to be the focus of care services and be actively engaged and empowered to manage their care, with the support of health care providers. We believe that health system efficiency, care quality and patient safety can be enhanced through the use of innovative, integrated, interactive, pro-active and personalized point-of- care solutions targeting both providers and patients. This is the premise for the IMPACT-AF study.

Primary care providers and their patients are anticipated to benefit from enhanced use of health information technology regarding the management of patients with AF. A clinical guideline-based decision support system (CDSS) will be developed and tested in primary care settings across Nova Scotia.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years (no max age limit)
* Confirmed atrial fibrillation.
* Able to provide informed consent in English.

Exclusion Criteria:

* Patients unable to provide informed consent.
* Patients who are not expected to be alive at the end of the 12 month follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1145 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jafna L Cox, MD, FRCPC, FACC, Principal Investigator — CDHA; Syed Sibte Raza Abidi, MSc, PhD, Study Director — Dalhousie University
Locations (2):
- Canada (2):
  - Capital District Health Authority, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not available due to ethics regulations.

REFERENCES:
- [Derived] Hamlin J, Cox J, Hamilton L, Nemis-White J, McKillop J, Sandila N, Parkash R. Regional Disparities in Atrial Fibrillation Management: An IMPACT-AF Substudy. CJC Open. 2024 Jul 3;6(10):1162-1169. doi: 10.1016/j.cjco.2024.06.010. eCollection 2024 Oct. PMID 39525336
- [Derived] Cox J, Hamilton L, Thabane L, Foster G, MacKillop J, Xie F, Ciaccia A, Choudhri S, Nemis-White J, Parkash R; IMPACT-AF Investigators. Computerized clinical decision support to improve stroke prevention therapy in primary care management of atrial fibrillation: a cluster randomized trial. Am Heart J. 2024 Jul;273:102-110. doi: 10.1016/j.ahj.2024.04.016. Epub 2024 Apr 28. PMID 38685464
- [Derived] Humphries B, Cox JL, Parkash R, Thabane L, Foster GA, MacKillop J, Nemis-White J, Hamilton L, Ciaccia A, Choudhri SH, Kovic B, Xie F. Resource use and cost associated with computerized decision support system and usual care in managing patients with atrial fibrillation: analysis of IMPACT-AF randomized trial data. BMC Med Inform Decis Mak. 2023 Oct 18;23(1):228. doi: 10.1186/s12911-023-02329-7. PMID 37853351
- [Derived] Nemis-White JM, Hamilton LM, Shaw S, MacKillop JH, Parkash R, Choudhri SH, Ciaccia A, Xie F, Thabane L, Cox JL; IMPACT-AF Investigators. Lessons learned from Integrated Management Program Advancing Community Treatment of Atrial Fibrillation (IMPACT-AF): a pragmatic clinical trial of computerized decision support in primary care. Trials. 2021 Aug 11;22(1):531. doi: 10.1186/s13063-021-05488-y. PMID 34380542
- [Derived] Humphries B, Cox JL, Parkash R, Thabane L, Foster GA, MacKillop J, Nemis-White J, Hamilton L, Ciaccia A, Choudhri SH, Xie F; IMPACT-AF Investigators. Patient-Reported Outcomes and Patient-Reported Experience of Patients With Atrial Fibrillation in the IMPACT-AF Clinical Trial. J Am Heart Assoc. 2021 Aug 3;10(15):e019783. doi: 10.1161/JAHA.120.019783. Epub 2021 Jul 28. PMID 34315232
- [Derived] Cox JL, Parkash R, Abidi SS, Thabane L, Xie F, MacKillop J, Abidi SR, Ciaccia A, Choudhri SH, Abusharekh A, Nemis-White J; IMPACT-AF Investigators. Optimizing primary care management of atrial fibrillation: The rationale and methods of the Integrated Management Program Advancing Community Treatment of Atrial Fibrillation (IMPACT-AF) study. Am Heart J. 2018 Jul;201:149-157. doi: 10.1016/j.ahj.2018.04.008. Epub 2018 Apr 7. PMID 29807323

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant did not meet inclusion criteria and was excluded from the analysis.
Groups:
- Clinical Decision Support System for AF: Providers randomized to access use of the Clinical Decision Support System (CDSS, a web-based tool).
  Clinical Decision Support System for AF: A web-based clinical decision support system, computerizing the Canadian AF clinical guidelines and best-practice approaches, to support primary care providers and patients in optimizing and standardizing AF care.
Period: Overall Study
Arm/Group | Clinical Decision Support System for AF | Usual Care
Started | 597 | 548
Completed | 590 | 543
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 7 | 4
Not completed — No baseline data | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Decision Support System for AF | Usual Care | Total
Number analyzed (Participants) | 590 | 543 | 1133
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (10.1) | 72.1 (9.9) | 72.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239 | 193 | 432
  Male | 351 | 350 | 701
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 329 | 308 | 637
  Ethnicity: Unknown | 216 | 200 | 416
  Ethnicity: Other | 45 | 35 | 80
Region of Enrollment [Count of Participants; unit: Participants]
  Canada: Rural Care Nova Scotia | 315 | 298 | 613
  Canada: Urban Care Nova Scotia | 275 | 245 | 520

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiovascular Hospitalization and AF-related Emergency Department Visits
Description: Any unplanned hospitalization (admission with an overnight stay in hospital) due to one of the following causes: acute coronary syndrome, pre-syncope /syncope, transient ischemic attack/ stroke, atrial fibrillation, flutter, pulmonary embolism /deep vein thrombosis /systemic embolism, worsening congestive heart failure including pulmonary edema or dyspnea of cardiac origin. AF-related ED visit was predefined as: any presentation with palpitations, rapid heart rate, presyncope or syncope, shortness of breath, transient chest discomfort, or hemodynamic instability resolving with cardioversion or rate-control, not resulting in hospitalization.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support System for AF | Usual Care
Number analyzed (Participants) | 590 | 543
Participants | 118 | 130

2. Secondary Outcome: Number of Participants With AF-related Emergency Department Visits
Description: * Individual element of primary outcome.
  * AF-related emergency department visits.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support System for AF | Usual Care
Number analyzed (Participants) | 590 | 543
Participants | 78 | 96

3. Secondary Outcome: Process of Care
Description: * Timely access to specialist consultation
  * Timely access to echocardiograms
  * Timely access to catheter ablations for AF and atrial flutter
Time Frame: 12 months
Population: Data were not available/collected from primary care provider charts that would permit analysis of the time between dates of referral and dates of access for the process of care outcomes.
Arm/Group | Clinical Decision Support System for AF | Usual Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Health Related Quality of Life
Description: - Health Related Quality of Life measured using an accepted health questionnaire (EQ-5D-5L).
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2021-06

5. Secondary Outcome: Costs
Description: * The costs associated with the development, implementation, and maintenance of CDSS.
  * The costs associated with managing and treating patients with AF.
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2021-09

6. Secondary Outcome: Cost Effectiveness
Description: - Incremental cost effectiveness ratio between the interventional arm and the control arm
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2021-09

7. Secondary Outcome: Number of Participations With CV Hospitalizations
Description: * Individual element of primary outcome.
  * AF-related emergency department visits.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support System for AF | Usual Care
Number analyzed (Participants) | 590 | 543
Participants | 40 | 26

8. Other Pre Specified Outcome: Number of Participants With Major Bleeding
Description: Major bleeding, as listed above, is to be defined as fatal bleeding and/or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome and /or overt bleeding causing a fall in hemoglobin level of 20 g/L or more, or leading to transfusion of two or more units of whole blood or red cells.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Decision Support System for AF | Usual Care
Number analyzed (Participants) | 590 | 543
Participants | 9 | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 12 months for each participant's active study phase.
Description: Safety outcomes were monitored and reported at 12 months, including Major bleeding per ISTH criteria as well as All bleeding.
Arm/Group | Clinical Decision Support System for AF | Usual Care
All-Cause Mortality (participants affected / at risk) | 28/590 | 21/543
Serious Adverse Events (participants affected / at risk) | 9/590 | 7/543
Other Adverse Events (participants affected / at risk) | 0/590 | 0/543
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Decision Support System for AF (N=590) | Usual Care (N=543)
Major bleeding per ISTH criteria (Vascular disorders) | 9 (9) | 7 (7)

LIMITATIONS AND CAVEATS:
Limitations can be found in the main outcomes paper, which is open access: https://www.sciencedirect.com/science/article/pii/S0002870320300855 The methods paper is also open access: https://www.sciencedirect.com/science/article/pii/S0002870318301170

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT01927367/SAP_000.pdf
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT01927367/Prot_001.pdf